CLINICAL TRIAL: NCT06660810
Title: Neoadjuvant Intralesional Injection of Talimogene Laherparepvec With Concurrent Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas
Brief Title: Neoadjuvant Intralesional Injection of Talimogene Laherparepvec
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Rieth (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, John Rieth, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202402722
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma; Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — talimogene laherparepvec; Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Expansion Pilot (Experimental): Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery. Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care
  Interventions: Drug: Talimogene Laherparepvec; Radiation: Neoadjuvant Radiation; Procedure: Surgery

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene laherparepvec (HSV-1 [strain JS1]/ICP34.5-/ICP47-/hGM-CSF) is an oncolytic immunotherapy, formerly known as OncoVEXGM-CSF, an immune-enhanced, oncolytic herpes simplex virus type 1 (HSV-1)
  Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec
Radiation: Neoadjuvant Radiation — Treatment given as a first step to shrink a tumor before the main treatment, which is usually surgery, is given.
  Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec
Procedure: Surgery — Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care

SUMMARY:
The proposed study is designed to treat locally advanced soft tissue sarcoma (STS) subtypes with neoadjuvant talimogene laherparepvec (TVEC) and preoperative external beam radiation therapy (EBRT).

DETAILED DESCRIPTION:
This is a single-arm open-label phase Ib and phase II clinical study assessing the safety and relative efficacy of concurrent talimogene laherparepvec in combination with radiotherapy in patients with soft tissue sarcomas. Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery. Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care.

ELIGIBILITY:
1. Subject has provided informed consent.
2. Histologically confirmed diagnosis of locally advanced STS subtypes (including undifferentiated pleomorphic sarcoma, myxofibrosarcoma, and malignant peripheral nerve sheath tumor (MPNST)) that are unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate.

   EXAMPLES:
   * Resectable stage IIB, III, and IV disease that are not suitable for surgical resection alone due to inability to achieve clear margins.
   * Including metastatic (stage IV) disease for which radiotherapy and surgical resection are indicated.
   * Sarcoma histologies to include: undifferentiated pleomorphic sarcoma (including the terms including, but not limited to pleomorphic undifferentiated sarcoma, unclassified spindle cell sarcoma, spindle cell sarcoma not otherwise specified, pleomorphic spindle cell sarcoma, pleomorphic fibroblastic sarcoma, undifferentiated high-grade pleomorphic sarcoma, pleomorphic sarcoma with prominent inflammation, pleomorphic sarcoma with giant cells, malignant fibrous histiocytoma fibrosarcoma), fibromyxosarcoma, and MPNST
3. Previous treatment: prior systemic anti-cancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy are allowed provided therapy completed at least1 year prior to enrollment.

   * No prior Talimogene laherparepvec or tumor vaccines allowed.
   * No prior radiation to the same tumor bed allowed.
4. Age ≥18 years.
5. Both men and women of all races and ethnic groups are eligible for this trial.
6. ECOG performance status ≤1.
7. Patient must have measurable disease:

   •Tumor size at least ≥ 5 cm in the longest diameter as measured by CT scan or MRI for which radiation is feasible.
8. Patient must have injectable disease (direct injection or ultrasound guided).

5.2 Eligibility Exclusion Criteria

1. Sarcoma histologies that are not consistent with undifferentiated pleomorphic sarcoma, myxofibrosarcoma, or MPNST
2. History or evidence of sarcoma associated with immunodeficiency states (e.g.:Hereditary immune deficiency, HIV, organ transplant or leukemia).
3. Subjects with retroperitoneal and visceral sarcoma.
4. History or evidence of uncontrolled gastrointestinal inflammatory bowel disease (ulcerative colitis or Crohn's disease) or other symptomatic uncontrolled autoimmune disease including, inflammatory bowel disease, or history of any poorly controlled or severe systemic autoimmune disease (i.e., severe rheumatoid arthritis requiring biologic treatment, systemic lupus erythematosus, scleroderma, or autoimmune vasculitis).

   History of other malignancy within the past 3 years except treated with curative intent and no known active disease present and has not received chemotherapy for ≥ 1 year before enrollment/randomization and low risk for recurrence.
5. History of prior or current splenectomy or splenic irradiation.
6. Active herpetic skin lesions
7. Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use.
8. Any non-oncology vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period.
9. Concomitant treatment with therapeutic anticoagulants such as warfarin. Patients on therapeutic low molecular weight heparin may be allowed provided the dose can be safely held as per the treating investigator on the morning of scheduled intratumoral injection and can be resumed 12 hours after the procedure.
10. Known human immunodeficiency virus (HIV) disease (requires negative test for clinically suspected HIV infection).
11. Acute or chronic hepatitis B or hepatitis C infection (requires negative test for clinically suspected hepatitis B or hepatitis C infection).

    * Evidence of hepatitis B -

      1. Positive HBV surface antigen (indicative for chronic hepatitis B or recent acute hepatitis B).
      2. Negative HBV surface antigen but positive HBV total core antibody (indicative for resolved hepatitis B infection or occult hepatitis B) and detectable copies of HBV DNA by PCR (detectable HBV DNA copies suggest occult hepatitis B).
    * Evidence of hepatitis C - a)Positive HCV antibody and positive HCV RNA by PCR (undetectable RNA copies suggest past and resolved hepatitis C infection).
12. Female subjects who are pregnant or breast-feeding or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment.
13. Female subjects of childbearing potential or male subjects who are unwilling to use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment. See Section 8.5 for more details.
14. Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
15. Other investigational procedures while participating in this study that could affect the primary objective of the study as determined by the PI are excluded
16. Subject previously has entered this study.
17. Evidence of CNS metastases.
18. History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec.
19. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
20. Patients on or requiring immunosuppressive therapies.
21. Any of the following laboratory abnormalities:

    * Hemoglobin < 9.0 g/dL
    * Absolute neutrophil count (ANC) < 1500 per mm3
    * Platelet count < 100,000 per mm3
    * Total bilirubin > 1.5 × ULN
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN
    * Alkaline phosphatase > 2.5 × ULN
    * PT (or INR) and PTT (or aPTT) > 1.5 × ULN
    * Creatinine > 2.0 × ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2030-03-10 (Estimated)

PRIMARY OUTCOMES:
pCR rate defined as the proportion of subjects with pathologic necrosis ≥ 90% | Weeks 12-14

SECONDARY OUTCOMES:
Adverse Events will be evaluated according to CTCAE version 4.0 | Initiation of treatment through Week 16
ORR defined as the proportion of subjects with a complete or partial response | Initiation of treatment through Week 12
TTP defined as time from first day of study treatment to first documented disease progression | Initiation of treatment through Week 12
Overall Survival defined as time from first day of study treatment to death due to any cause | Initiation of treatment through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States